CLINICAL TRIAL: NCT03226158
Title: Prediction of Adverse Events in Children and Adolescents With Cancer at High Risk of Infection (PREDSEQ)
Brief Title: Next Generation Pathogen Sequencing for Prediction of Adverse Events
Status: Active, not recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Karius, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PREDSEQ
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Bloodstream Infection
Keywords: Next generation pathogen sequencing (NGPS); Pediatric; Cancer; Bloodstream infection (BSI)
MeSH Terms: conditions — Sepsis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples collected but not required for clinical care will undergo next generation pathogen sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The majority of children and adolescents diagnosed with cancer will experience one or more episodes of fever or infection during their course of therapy. The most common microbiologically documented infection is bloodstream infection (BSI), which can be associated with severe sepsis or death. Current methods of diagnosis require a significant load of live bacteria in the blood making early detection difficult. Delayed diagnosis and delayed optimal therapy of BSIs are associated with increased morbidity and mortality.

This study seeks to identify whether next generation sequencing (NGS) of pathogens can identify patients with impending bloodstream infection. This would enable preemptive targeted therapy to replace antibacterial prophylaxis which often leads ot high-density broad-spectrum antibiotic exposure and contributes to subsequent development of antibiotic resistance.

PRIMARY OBJECTIVE:

* To estimate the sensitivity and specificity of next generation pathogen sequencing for prediction of bloodstream infection in children with cancer at high risk of infection.

DETAILED DESCRIPTION:
Plasma samples collected but not required for clinical care (discarded samples) will be collected and stored. Results of NGS will be compared between patients who develop BSI immediately (within 72 hours) after sample collection, those who develop other infectious syndromes, and those who remain well. Clinical data describing baseline information about the patient and malignancy, antibiotic and chemotherapy exposure, microbiology testing, hematology results, and infection-related events will be collected prospectively from the electronic medical record.

An initial exploratory phase will examine approximately 50 participants to determine whether the effectiveness of predicting infections. The study may then enroll up to 200 participants to collection additional data for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Under 25 years of age at time of study enrollment
* Undergoing care for cancer at St. Jude
* In a category of patients who are considered by the investigator to be at high risk of infection
* Expected to receive care at St. Jude for at least 7 days

Exclusion Criteria:

* Any condition that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants who are being treated at St. Jude Children's Research Hospital and who have a high risk of infection.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of NGS-positive results | Once (within 72 hours of enrollment)
  To estimate the sensitivity of next generation pathogen sequencing for prediction of BSI, the proportion of NGS-positive results in all positive BSI cultures will be given.
Proportion of NGS-negative results | Once (within 72 hours of enrollment)
  To estimate the specificity of next generation pathogen sequencing for prediction of BSI, the proportion of NGS-negative results in all negative BSI cultures will be given.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Wolf, MBBS, BA, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Goggin KP, Gonzalez-Pena V, Inaba Y, Allison KJ, Hong DK, Ahmed AA, Hollemon D, Natarajan S, Mahmud O, Kuenzinger W, Youssef S, Brenner A, Maron G, Choi J, Rubnitz JE, Sun Y, Tang L, Wolf J, Gawad C. Evaluation of Plasma Microbial Cell-Free DNA Sequencing to Predict Bloodstream Infection in Pediatric Patients With Relapsed or Refractory Cancer. JAMA Oncol. 2020 Apr 1;6(4):552-556. doi: 10.1001/jamaoncol.2019.4120. PMID 31855231
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols